CLINICAL TRIAL: NCT05422040
Title: Effectiveness of Diathermy Compared to Dry Needling in the Short-term Management of Subjects With Chronic Low Back Pain: a Randomised Controlled Trial
Brief Title: Dry Needlig Vesus Tecartherapy in Low-back Pain Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIM/HU/2019/30
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Low Back Pain
Keywords: Back pain, dry needling, Tecartherapy
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): Dry needling is performed with a 4cm needle (APS Dry Needles®) on the most symptomatic side of the patient on palpation. To perform the technique, the patient is positioned in prone position on the couch. The physiotherapist palpates the lateral border of the lumbar iliocostalis muscle and performs the tapping technique in a latero-medial direction parallel to the stretcher.
  The technique is performed by applying 12 incisions. After the application of the technique, ischaemic compression shall be performed for 1 minute.
  Patients will complete a home exercise program
  Interventions: Other: Dry needling
- Diathermy treatment (Experimental): Diathermy treatment will be applied using the TCaRe Power diathermy instrument (PRIM Physio©), using a capacitive system with an intensity of 50%, with slight variation depending on patient tolerance and 500khz. The therapy will be applied for 10 minutes on each side of the patient's lumbar region, who will be positioned in prone decubitus during the intervention.
  Patients will complete a home exercise program
  Interventions: Other: Tecartherapy treatment

INTERVENTIONS:
Other: Dry needling — Invasive treatment will be performed on the most symptomatic lumbar iliocostalis muscle.
  Arms: Dry needling
Other: Tecartherapy treatment — Treatment will be carried out with deep thermotherapy in the lumbar region.
  Arms: Diathermy treatment

SUMMARY:
Introduction: Diathermy is a new tool that could help subjects with chronic low back pain (CLBP), with no studies having compared it to other interventions already investigated such as dry needling.

Hypothesis: Diathermy is more effective than dry needling in improving pain intensity in the short term in subjects with CLBP.

Design: randomised controlled trial Methods: We will conduct a convenience sampling, with subjects receiving 2 treatment sessions with diathermy or dry needling, according to allocation. Subjects will be assessed at baseline, 1 week, 1 month and 3 months after treatment for pain intensity, disability, kinesiophobia and catastrophizing. Analysis of variance (ANOVA) and moderation analysis will be performed to evaluate the results, with 95% confidence intervals (CI).

DETAILED DESCRIPTION:
A prospective longitudinal experimental randomised controlled trial study will be conducted from August 2022 to March 2023. The study will be conducted in accordance with the recommendations of the Consolidated Standards of Reporting Trials (CONSORT) statement,15 and in accordance with the Declaration of Helsinki.

Subjects were randomly assigned to one of the two intervention groups:

Diathermy. Diathermy treatment was applied using the TCaRe Power diathermy instrument (PRIM Physio©), using a capacitive system with an intensity of 50%, with slight variation depending on patient tolerance and 500khz. The therapy will be applied for 10 minutes on each side of the patient's lumbar region, who will be positioned in prone decubitus during the intervention.

The application will be active along with massage techniques. Dry needling. Dry needling is performed with a 4cm needle (APS Dry Needles®) on the most symptomatic side of the patient on palpation. To perform the technique, the patient is positioned in prone position on the couch. The physiotherapist palpates the lateral border of the lumbar iliocostalis muscle and performs the tapping technique in a latero-medial direction parallel to the stretcher.

The technique is performed by applying 12 incisions. After the application of the technique, ischaemic compression shall be performed for 1 minute.

Patients will complete a home exercise program

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Chronic non-specific low back pain.
* Duration of pain of more than 6 weeks.

Exclusion Criteria:

* Neurological signs or symptoms.
* Radicular pain.
* Radiating pain below the knee.
* Belonephobia.
* Traumatic processes and/or surgeries in the lumbar region in the last year.
* Having received physiotherapy treatment in the last 3 months.
* Systemic diseases such as cancer, rheumatic diseases, neurological diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | Change from baseline at 3 months
  The visual analogue scale (VAS) is a 10cm long line where 0 indicates no pain at all and 10 the worst pain imaginable. It is a tool that has shown good reliability values (r = 0.94).

SECONDARY OUTCOMES:
Rolland-Morris questionnaire | Change from baseline at 3 months
  The questionnaire scores from 0 (no disability) to 24 (maximum degree of disability), its cross-cultural adaptation to Spanish has shown good concurrent validity values (r = 0.34-0.57) and good reliability values (Intraclass Correlation Coefficient = 0.87).
Tampa Scale for Kinesiophobia 11 (TSK-11) | Change from baseline at 3 months
  The questionnaire is scored from 11 to 44, the score being represented as a percentage from 0% (minimum degree of kinesiophobia) to 100% (maximum degree of kinesiophobia). The cross-cultural adaptation of the TSK-11 to Spanish has shown good concurrent validity values (r = 0.27-0.49) and good reliability values (r = 0.55).
Pain Catastrophism Scale | Change from baseline at 3 months
  The questionnaire is scored from 0 to 54 and is represented as a percentage from 0% (minimum degree of catastrophism) to 100% (maximum degree of catastrophism). The cross-cultural adaptation to Spanish has shown good values of concurrent validity (r = 0.28-0.66) and reliability (Intraclass Correlation Coefficient = 0.84).
Pressure pain threshold | Change from baseline at 3 months
  The pressure pain threshold (PPT) will be measured using a hand-held algometer (Wagner Force Dial, Model FDK 20, Wargner Instruments, Greenwich, CT, USA). This algometer has a 1cm2 surface area tip that records the pressure in kg/cm2. The algometer has been shown to be a valid and reliable tool for the measurement of UDP, with Intraclass Correlation Coefficient values in subjects with low back pain of 0.93.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pecos-Martín, PhD, Principal Investigator — Alcala University
Locations (1):
- Centro Investigación Fisioterapia y Dolor, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No